CLINICAL TRIAL: NCT06941220
Title: Effect of Mulligan Versus Maitland Mobilization on Lumbar Proprioception in Patients With Chronic Nonspecific Low Back Pain
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator : alshaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005680
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain
Keywords: mulligan; maitland; proprioception; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: mulligan and maitland parallel group
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mulligan group (Experimental): thirty patients will receive mulligan sustained natural apophyseal glide (SNAG) for each level was 3 sets of 6 repetitions 3 times per week for 1 month plus traditional therapy
  Interventions: Other: mulligan group; Other: traditional therapy
- Maitland mobilization (Experimental): thirty patients will receive Maitland 3 times per week for 1 month plus traditional therapy
  Interventions: Other: Maitland mobilization; Other: traditional therapy
- traditional therapy (Active Comparator): thirty patients will receive traditional therapy three times a week for four weeks
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: mulligan group — SNAG technique was applied from a sitting position on the edge of the table while both feet were on a foot rest. A specialized Mulligan belt was used around the patient's waist and therapist's hips. The mobilizing force was applied parallel to the facet joint plane (cephalic direction) and over the spinous processes of the respective symptomatic spinal levels. The patients were asked to lean forward as much as possible during application of the mobilizing force and then return to the starting position while the therapist maintained his mobilizing force until the end. plus traditional therapy
  Arms: mulligan group
Other: Maitland mobilization — The subjects were placed in the prone position on a plinth with their hands beside them, and the therapist stood on the subject's side, the ulnar surface of the hand (between pisiform and hamate) was placed over the hypomobile spinous process. The second hand was placed on top of the first to enhance its force. With the therapist's elbows slightly bent and shoulders exactly above the spinous process, an oscillatory movement of the vertebra was executed by applying a posterior-anterior force to the hypomobile or painful spinous process.
  Grade III mobilization was applied four times, each with 60 s of oscillation and 20 s of rest in between them (2 or 3 oscillations per second) plus traditional therapy
  Arms: Maitland mobilization
Other: traditional therapy — the patients will receive traditional therapy in the form of passive stretching, strengthening, and lumbar stabilization exercises

SUMMARY:
this study will be conducted to compare between the effect of mulligan mobilization versus Maitland mobilization on pain ,function and lumbar proprioception in patients with chronic nonspecific low pain

DETAILED DESCRIPTION:
Low back pain (LBP) is considered as one of the most widespread musculoskeletal disorders, impacting over 80% of the world's population, resulting in work absence, medical consultation, a decline in quality of life, and financial burden. Lumbar repositioning error was high around 30° of trunk flexion in individuals with CLB. When lumbar proprioceptive deficiencies arise, the activation pattern of back muscles is disturbed, the mechanics of the spinal unit differs from that of a healthy spine, and the recurrence rate of LBP increases . CLBP is managed using various intervention modalities, including drug therapy and physical therapy approaches . Physical therapy modalities, such as manual therapy, therapeutic exercises, and biopsychosocial techniques, are used for treating LBP. Manual therapy is a common and suggested modality for treating CLBP that has strong evidence. It is employed in physical therapy practice, including Maitland mobilization and Mulligan mobilization. Mulligan mobilization as well as Maitland mobilization has significant effect on pain ,function disability and lumbar repositioning error. But there is gap about which is more beneficial. So we conduct this study to determine which technique is more beneficial for patients

ELIGIBILITY:
Inclusion Criteria:

* They had interrupted or continuous LBP symptoms for more than 3 months
* both gender

Exclusion Criteria:

* specific LBP
* those who were pregnant
* those with neurological problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
joint position error (lumbar proprioception) | up to four weeks
  joint position error will be measured by isokinetic. The lumbar Joint Position Error (JPE) Test is a measurement tool used to clinically assess an individual's lumbarcephalic proprioception ability. proprioception describes one's sense of position of their back in space. The lumbar JPE Test measures the ability of a blindfolded patient to accurately relocate their lumbar to a predetermined neutral point after lumbar joint movement.

SECONDARY OUTCOMES:
pain intensity | up to four weeks
  pain intensity will be measured by VAS. The VAS is a 10-cm horizontal line and has two ends-one end expresses no pain on the left side and the second end expresses maximal pain on the right side
Functional disability | up to four weeks
  The Arabic version of the Oswestry Disability Index (ODI) was used to assess functional level. The ODI is a 10-item questionnaire, with each item answered using a 6-point Likert scale, ranging from 0 to 5. Pain severity, self-care, sitting, lifting, sleeping, walking, traveling, sexual life (if founded), and sociality are all items considered by the ODI.The point total from each section is summed, divided by the total points possible of all sections answered, and multiplied by 100 to create a percentage disability from 0-100%, with a lower percentage indicating less disability.
lumbar range of motion | up to four weeks
  range of motion will be measured by tape measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Alshaymaa Shaaban Abdelazeim, Giza, Doki, Egypt